CLINICAL TRIAL: NCT02265653
Title: Randomised 3-way Cross-over Phase I Study to Investigate the Relative Bioavailability of BIIL 284 BS 75 mg Tablet C and Tablet D in Comparison to WIF Tablet in Healthy Volunteers
Brief Title: Relative Bioavailability, Pharmacokinetics, Safety and Tolerability of BIIL 284 BS in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 543.3
Record Dates: First submitted 2014-10-15; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (3):
- BIIL 284 BS tablet C (Experimental)
  Interventions: Drug: BIIL 284 BS tablet C
- BIIL 284 BS tablet D (Experimental)
  Interventions: Drug: BIIL 284 BS tablet D
- BIIL 284 BS WIF tablet (Active Comparator)
  Interventions: Drug: BIIL 284 BS WIF tablet

INTERVENTIONS:
Drug: BIIL 284 BS tablet C
  Arms: BIIL 284 BS tablet C
Drug: BIIL 284 BS tablet D
  Arms: BIIL 284 BS tablet D
Drug: BIIL 284 BS WIF tablet
  Arms: BIIL 284 BS WIF tablet

SUMMARY:
The objective of the present study is to investigate the relative bioavailability of two BIIL 284 BS tablets (tablet C and tablet C) in comparison to the WIF tablet at a dose of 75 mg following a standard breakfast in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* All participants are healthy males
* Age range from 21 to 50 years
* Broca-Index: within +- 20% of their normal weight
* In accordance with Good Clinical Practice (GCP) and local legislation each volunteer is supposed to give their written informed consent prior to admission to the study

Exclusion Criteria:

* Volunteers will be excluded from the study if the results of the medical examination or laboratory tests are judged by the clinical investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* Volunteers with history of orthostatic hypotension, fainting spells or blackouts
* Volunteers with chronic or relevant acute infections
* Volunteers with history of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Volunteers who have taken a drug with a long half-life (>= 24 hours) within one month or less than ten half-lives of the respective drug before enrollment in the study
* Volunteers who received any drugs which might influence the results of the trial the week previous to the start of the study
* Volunteers who participated in another study with an investigational drug within the last two months preceding this study
* Volunteers who smoke (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Volunteers who drink more than 60g of alcohol per day
* Volunteers who are dependent on drugs
* Volunteers who participated in excessive physical activities (e.g. competitive sports) within the last week before the study
* Volunteers who have donated blood within the last 4 weeks (>= 100 mL)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1999-11; Primary Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 72 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRTtot (Total mean residence time) | up to 72 hours after drug administration
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 72 hours after drug administration
CLtot/F (Total clearance after oral administration) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with clinically findings in vital functions | up to 8 days after last drug administration
  blood pressure, pulse rate, ECG
Number of subjects with clinically findings in laboratory tests | up to 8 days after last drug administration